CLINICAL TRIAL: NCT03776448
Title: The Effect of 2 Grams Daily Supplementation of Thymoquinone -Containing Sativa Nigra Oil on Blood Glucose Levels of Adults: A Placebo-controlled Double-blinded Randomized Controlled Trial
Brief Title: The Effect of 2 Grams Daily Supplementation of Sativa Nigra Oil on Blood Glucose Levels of Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sulaiman AlRajhi Colleges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SulimanAC-BlackseedOil
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participants and researchers involved directly in collecting data (ex. Measuring blood pressure or interviewing subjects) will be unaware of the allocation status and thus blinded. However, statistical analysts and those who will provide the participants with the intervention/placebo will be aware of the allocation status. All interventions (black seed oil and charcoal softgels) will be supplemented in neutral identical containers. Each participant will receive a container labeled with his or her specific identification code and containing the intervention for the arm to which he or she has been allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sativa Nigra oil arm (Experimental): A total of 15 subjects randomly allocated to the treatment arm will receive 2000mg a day of 'Sativa Nigra oil' softgels for 30 consecutive days. The total daily dose is divided in 4 doses taken 6 hourly (each softgel contains 500mg). This supplement is manufactured by [Bioextract Ltd, Sri Lanka] and is available commercially.
  Interventions: Dietary Supplement: Sativa Nigra oil Softgels
- The charcoal arm (Placebo Comparator): Subject randomly allocated to the control arm will receive 1040mg a day of activated charcoal softgels for 30 consecutive days. The total daily dosage is divided in 4 doses taken 6 hourly (each softgel contains 260mg). This supplement is manufactured by [Arkopharma Pharmaceutical Laboratories] and is available commercially.
  Interventions: Dietary Supplement: Activated Charcoal Softgels

INTERVENTIONS:
Dietary Supplement: Sativa Nigra oil Softgels — Nigella sativa, a flowering plant native to southwest Asia, is considered one of the most important healing medicinal plants in Islamic culture. The use of its richly colored black seeds has been recommended in the prophetic medicine. It's also known by various other names amongst different cultures. Importantly, its seed is known in Arabic as 'habat al Baraka' which translates literally to 'the seed of blessing'.The active ingredient is believed to be thymoquinone richly present in the oil extract of its seeds. Apart from mild occasional gastrointestinal disturbance, black seed oil has no side effects and is considered very safe. .
  Other Names: Blackseed oil softgels
  Arms: Sativa Nigra oil arm
Dietary Supplement: Activated Charcoal Softgels — This supplement is manufactured by [Arkopharma Pharmaceutical Laboratories] and is available commercially. The use of activated charcoal softgels as a placebo is documented in several other clinical trials. The single most relevant characteristic of charcoal is its minimal if any gastrointestinal absorption. As a result, it does not undergo any metabolism and is excreted completely in feces. This makes charcoal an attractive placebo choice for small trials or when manufacturing a specific placebo is not feasible. Charcoal softgels are black in color and resemble black seed oil softgels to a great extent.
  Arms: The charcoal arm

SUMMARY:
Diabetes mellitus is a growing global concern with significant health and financial burdens. The Kingdom of Saudi Arabia is one of the world's top 10 countries with the highest diabetes prevalence. Strict blood glucose control is an important measure in the treatment of diabetes and prevention of its complications. The scientific community has recently shown a profound interest in the area of complementary and alternative medicine where a ton of research is being conducted. The primary focus of this field of research is subjecting many of the medicinal plants used in herbalism to the scientific methodology of testing. In order for these plants to be implemented in treatment protocols, their effect must be clearly proven and documented scientifically. This study aims to investigate the effect of daily consumption of black seed oil on the blood sugar levels of healthy adults.

DETAILED DESCRIPTION:
1. Research Question and Objectives:

   Research question: Will daily consumption of 2g of N. sativa extract oil improve (decrease) fasting blood glucose levels of adults?

   Research Objectives:

   Primary: To conduct a feasibility study investigating the effect of daily consumption of 2g of N. sativa extract oil on the fasting blood glucose levels of adults.

   Secondary: To investigate the effect of daily consumption of 2g of N. sativa oil extract on blood pressure.

   Secondary: To investigate the feasibility of regular black seed oil intake by means of gastrointestinal symptoms questionnaire
2. Trial Design:

   Design: This is a placebo-controlled double-blinded randomized controlled trial with two parallel groups.

   Allocation: The randomization will substantially reduce the risk of selection bias and confounding factors. Simple randomization will be used in this study. This randomization will insure a balanced 1:1 allocation ratio at the end of sample recruitment. A computer program will be used to generate a set of random numbers, an allocation sequence. Each number assigns the participant either to the intervention or the control group. However, this information will only be revealed after a sealed opaque file is opened at the time of recruitment.

   Framework: Exploratory study to gather preliminary information on the intervention and the feasibility of its use in blood glucose control.
3. Study Setting:

   This study will be conducted in the internal clinics of Sulaiman Al Rajhi Colleges in Qassim region, Kingdom of Saudi Arabia.
4. Participants Timeline:

   The primary outcome (Fasting blood glucose, FBG) will be assessed three times during the study period. FBG measurement moments for each participant are at 0, 2, and 4 weeks from the time of randomization. The rationale behind spacing measuring moments two weekly is to allow a sufficient response time for FBG levels to be interpretable. Secondary outcomes will be assessed weekly totaling five assessments at 0, 1, 2, 3 and 4 weeks from the time of randomization. The participant will have to visit the College internal clinics at his or her respective measurement points. The participant will be reminded the night before to remain fasting for at least 6 hours before the visit. At each visit, the participant will initially answer a set of questions to assess the degree of compliance and adherence. He or she then will be asked to report any possible side effects and will be allowed a time to fill in the questionnaires and express any concerns he or she might have. Next, blood pressure will be measured. Finally, a venous blood sample will be taken to measure the fasting blood glucose.
5. Recruitment:

   The participants in this study are going to be recruited form Sulaiman Al Rajhi Colleges, Al-Qassim, Kingdom of Saudi Arabia. Multiple channels will be used to recruit subjects including but not limited to: invitation posters/flyers, E-mails and social media. Prospective participants will be subjected to our inclusion/exclusion criteria to determine their eligibility and finalize their recruitment and randomization. Each participant will have to provide a written informed consent in order be enrolled.
6. Data Collection:

Primary outcome: Trained personnel will be responsible for obtaining venous blood samples from all subjects in a controlled and private environment. Each sample will be labeled with the participant's unique identification code and sent immediately to a cooperating external lab equipped with advanced and accurate devices.

Secondary outcomes: Each participant will have his or her blood pressure measured privately in the internal clinic by trained personnel using a standardized sphygmomanometer. The side effects of the intervention will be assessed by means of a questionnaire specifically developed for the purpose. The use of a standardized questionnaire is not necessary since the data is not intended to diagnose or categorize any particular health condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-60
* Regular Student or Faculty in Sulaiman Alrajhi Colleges
* Consenting for intervention and follow up

Exclusion Criteria:

* Type I diabetes or Insulin Therapy
* Significant chronic medical illness
* Current use of long-term prescription drugs
* Current use of black seed oil
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Fasting venous blood glucose | The primary outcome will be assessed at 1 week, 2 weeks, 3 weeks and 4 weeks of intervention
  The change from baseline in fasting venous blood glucose after 1 month of intervention. The participant-level analysis is change from baseline at 1 month and the method of aggregation for each study group is the mean.

SECONDARY OUTCOMES:
Blood pressure | This outcome will be assessed at 1 week, 2 weeks, 3 weeks and 4 weeks of intervention
  the change from baseline in mean seated blood pressure after 1 month of intervention. The participant-level analysis is change from baseline at 1 month and the method of aggregation for each study group is the mean
Gastrointestinal symptoms | This outcome will be assessed at 1 week, 2 weeks, 3 weeks and 4 weeks of intervention
  The proportion of subjects reporting significant gastrointestinal symptoms defined as moderate or severe in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nazmus Saquib, Phd, Principal Investigator — SRC
Locations (1):
- Sulaiman AlRajhi Colleges, Al Bukairiyah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No